CLINICAL TRIAL: NCT06610565
Title: Fasting-mimicking Diet: A Randomized Trial on Feasibility, Safety and Effects of Multicycle Dietary Intervention on Side Effects of Aromatase Inhibitors Treatment in Post-menopausal Patients With Breast Cancer
Brief Title: Fasting-mimicking Diet Intervention on Side Effects of Aromatase Inhibitors Treatment in Patients With Breast Cancer
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: European Institute of Oncology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: IEO 1570
Record Dates: First submitted 2024-09-20; First posted 2024-09-24 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Breast Cancer
Keywords: fasting-mimicking diet
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Intervention Model Description: 1:1 randomization into two arms: one intervention, where will receive nutritional counseling and the study diet for 5 days each month for 6 months, and a control one, where they will receive only nutritional counseling.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention arm (Experimental): intervention arm where will receive nutritional counseling and the study diet for 5 days each month for 6 months
  Interventions: Dietary Supplement: FASTING-MIMICKING DIET PROGRAM
- control arm (Experimental): control arm where they will receive only nutritional counseling
  Interventions: Dietary Supplement: FASTING-MIMICKING DIET PROGRAM

INTERVENTIONS:
Dietary Supplement: FASTING-MIMICKING DIET PROGRAM — Nutritional intervention via fasting-mimicking diet. Patients receiving adjuvant therapy with aromatase inhibitors will be randomized 1:1 into two arms: one intervention, where will receive nutritional counseling and the study diet for 5 days each month for 6 months,and a control one, where they will receive only nutritional counseling.

SUMMARY:
The primary endpoint of this study is to determine whether cycles of short term FMD exposure to a fasting-mimicking diet is effective in reducing total cholesterol levels.

DETAILED DESCRIPTION:
the short term FMD exposure to a fasting-mimicking diet reduce total cholesterol levels

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* WHO performance status score 0-2
* Early stage breast cancer, ER positive, receiving an adjuvant endocrine treatment with aromatase inhibitor
* Hypercholesterolemic (total cholesterol >200mg/dL)
* Ongoing treatment with aromatase inhibitors (at least six months of drug exposure)
* Adequate renal, hepatic, and hematopoietic function
* Written and informed consent for biomaterial submission and participation in the clinical trial
* Compliance with treatment and follow up protocol
* No other investigational agent may be administered concurrently to patients enrolled in this trial
* Patients with skeletal pain are eligible if bone scan and/or RX examination fails to disclose metastatic disease
* The interval between the onset of systemic adjuvant therapy with AIs and the randomization should be at least 6 months
* Patient is accessible geographically for follow-up and must be able to provide dietary data via telephone recalls
* Must be medically able to accept either dietary supplementation group prior to randomization.

Exclusion Criteria:

* Underweight (BMI < 18.5 kg/m2)
* Current or past eating disorders identified with the SCOFF Questionnaire (Useful Eating Disorder screening questions) [19]
* Malnutrition Universal Screening Tool (MUST). It considers body mass index, weight change and acute disease effect equally and determines a malnutrition risk score. A score ≥1 identify a patient at moderate risk of malnutrition;
* Treatment with any investigational or non-registered drug other than the study product(s) within 30 days preceding the first dose of study product, or planned use during the study period
* Use of statins or supplements similar to statins (e.g red rice) or other drugs that interfere with lipid absorption (e.g ezetimibe)
* Known to have difficult-to-control hypertension, coronary artery disease, arrhythmia requiring treatment, clinically significant valvular disease, cardiomegaly on chest X-ray, ventricular hypertrophy on ECG, previous myocardial infarction, or congestive heart failure Patients with diabetes are not eligible for the study
* History of allergic reactions likely to be exacerbated by any component of the investigational product used in the study
* Other concurrent, severe medical problems, unrelated to the malignancy, that would significantly limit full compliance with the study or expose the patient to unacceptable risk
* Previous or concomitant malignancies at other sites, except effectively treated malignancy that is considered by the Investigator to have been cured
* Psychiatric or addictive disorders that may compromise the ability to give informed consent or to comply with study procedures.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — only female
Enrollment: 60 (Estimated)
Dates: Start 2024-09-01 (Actual); Primary Completion 2027-04-01 (Estimated); Study Completion 2027-04-01 (Estimated)

PRIMARY OUTCOMES:
Fasting-mimicking diet | from baseline to the end of treatment at 12 month
  Determination of number of cycles of short term FMD exposure to a fasting-mimicking diet in reducing total cholesterol levels

CONTACTS AND LOCATIONS:
Overall Officials: Giuseppe Curigliano, Principal Investigator — IEO
Locations (1):
- IEO, Milan, Italy, Italy